CLINICAL TRIAL: NCT02939547
Title: A Phase I Study to Evaluate the Single and Multiple-dose Pharmacokinetics of Intravenous Trappsol Cyclo (HP-Beta-CD) in Patients With Niemann-Pick Disease Type C (NPC-1) and the Effects of Dosing Upon Biomarkers of NPC Disease
Brief Title: Study of the Pharmacokinetics of Trappsol and Effects on Potential Biomarkers of Niemann-Pick C1 (NPC1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cyclo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: CTD-TCNPC-101
Record Dates: First submitted 2016-09-21; First posted 2016-10-20 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Niemann-Pick Disease, Type C1
Keywords: intravenous; cyclodextrin; compassionate; Trappsol
MeSH Terms: conditions — Niemann-Pick Disease, Type C | interventions — 2-Hydroxypropyl-beta-cyclodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hydroxypropyl-beta-cyclodextrin IV 1500 mg/kg (Active Comparator): Hydroxypropyl-beta-cyclodextrin administered by slow IV infusion for 8 - 9h every 2 weeks
  Interventions: Drug: Hydroxypropyl-beta-cyclodextrin
- Hydroxypropyl-beta-cyclodextrin IV 2500 mg/kg (Active Comparator): Hydroxypropyl-beta-cyclodextrin administered by slow IV infusion for 8 - 9h every 2 weeks
  Interventions: Drug: Hydroxypropyl-beta-cyclodextrin

INTERVENTIONS:
Drug: Hydroxypropyl-beta-cyclodextrin — Used in the treatment of Niemann-Pick Disease C1 ( NPC1)
  Other Names: Hydroxypropyl-beta-cyclodextrin (HP-β-CD)

SUMMARY:
This research study is being conducted to find out whether Trappsol® Cyclo™, an experimental treatment for people with Niemann Pick disease Type C (NPC-1) is safe at 2 different dose levels and what effects it has on people who have this condition. NPC-1 is caused by a defect in the protein which is important for the transport of fatty substances like cholesterol out of cells. Without this protein, fats build up in the cells ultimately leading to organ damage. The way in which this experimental treatment works is not fully understood but laboratory experiments have shown that it can potentially remove cholesterol build up from the cells in people who have NPC-1. Approximately 12 patients will be asked to take part in this research study for up to 20 weeks (w) in total (including screening. treatment and follow-up). Recruitment is expected to take 6- 9 months.Patients who take part will receive treatment by an intravenous infusion every two weeks. The study will look at what the body does to the drug as well as what the drug does to the body by taking and examining blood and urine samples. A sample(s) of cerebrospinal fluid (CSF) will be taken by lumbar puncture during the first treatment dose and may be collected during subsequent doses. Liver and skin biopsy specimens will be taken to assess filipin staining. Cholesterol metabolism will be investigated in liver samples and splenic and hepatic elasticity will be assessed by ultrasound. Patients will also have their hearing tested, be asked questions by their doctor as well completing questionnaires to help assess any changes in their condition during treatment.This study is being sponsored and funded by CTD holdings Inc. It is planned to be run in the USA,.

DETAILED DESCRIPTION:
The planned study has been designed as a Phase I, double-blind, randomised, multi-centre, parallel group study based on information and data available from the administration of Trappsol Cyclo via compassionate/named patient use in patients with NPC-1, and data on other cyclodextrin products in the scientific literature.

The study is comprised of a screening phase of up to 4w a treatment phase of 12w and a 4w follow-up. The primary objective is to compare the plasma pharmacokinetics of single and multiple doses of two different levels of IV Trappsol Cyclo. Secondary objectives include investigation of the HP-β-CD effect of different doses of IV Trappsol Cyclo upon serum and lymphocytic markers of cholesterol metabolism and evaluation of Trappsol concentrations in the cerebrospinal fluid (CSF) following IV administration , evaluation of the impact of treatment upon measures of neurological function including ataxia, aphasia and saccadic eye movements, and the impact of treatment upon behavioral aspects of NPC-1.

It is planned to recruit a total of 12 patients to the study. Patients will be randomised 1:1 to one of the two dose levels (1500 mg/kg or 2500 mg/kg; six patients per dose level). Treatment will be administered every two weeks by slow IV infusion over 8 to 9 hours at different concentrations to achieve the proscribed dose levels. Patients will receive treatment for a total of 12 weeks. Patients who withdraw prior to completion of the initial pharmacokinetic and pharmacodynamic assessments will be replaced.

The design of the proposed study thus enables early assessment of potential biochemical markers of response but allows for a sufficient dosing duration to enable the short-term effectiveness of Trappsol in NPC to be assessed.

The maximum dose proposed for this study is below the maximum dose for which long term clinical data is available in 2 patients (2800 mg/kg weekly for 3-5 years). Although individual clinicians have not always utilized an escalating rate of infusion, the reports of infusion related reactions in three patients suggest that this is an appropriate clinical strategy to mitigate the risk of such events and is consistent with dosing administration for other therapeutic agents. In the proposed study, treatment will be administered less frequently than has been undertaken in compassionate use. This longer dosing interval is supported by nonclinical data comparing the metabolism of cholesterol in non-human species with that in man; although a once weekly dosing interval was initially studied in man based on data in the mouse, HP-β-CD cholesterol metabolism/turnover in the mouse is 13-fold higher than in man which, in NPC, likely translates into a 13-fold slower accumulation of cholesterol in human cells compared with those of the mouse. Therefore, it is theorized that, given the slower cholesterol metabolism in humans, the dosing interval could be much less frequent in man than in mouse; however, based on what is known about cholesterol metabolism in humans and the pharmacokinetic and pharmacodynamic effect of HP-β-CD in the mouse, a dosing interval of 2 weeks in man is likely to be well within the therapeutic dosing interval and also minimizes the amount of infusions required to be administered.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of NPC-1 defined as one of the following

   1. Two NPC-1 mutations on exome gene sequencing
   2. One NPC-1 mutation and positive filipin staining (current or prior)
   3. Vertical supranuclear gaze palsy [VSGP] plus either ≥ one NPC-1 mutation or positive filipin staining and no NPC-2 mutations
2. NIH NPC Severity Score <30 and with no more than 4 individual domains with a score ≥ 3.
3. Age range: 18 years upwards
4. At least one systemic manifestation of NPC disease defined as one or more of

   1. Clinically detectable hepatomegaly and/or either ALT or AST outside the normal range for the study laboratory
   2. Clinically detectable splenomegaly
   3. Impaired respiratory function due to NPC or a history of pneumonia in the last 12 months
5. Negative urine pregnancy test for females of child bearing potential
6. Written, informed consent

Exclusion Criteria:

1. The presence of NPC-2 mutations on exome gene sequencing
2. Previous receipt of cyclodextrin therapy within 3 months of baseline
3. Receipt of any of the following medications within 1 month of baseline: Coenzyme Q10, curcumin, cinnamon, fish oil supplements, high dose vitamin D (>500 milli-International unit (mIU)/day), acetyl leucine, or gingko biloba
4. Concurrent treatment with any therapy indicated for the lowering of cholesterol such as statins, fibrates, ezetimibe
5. Karnofsky score < 40
6. Inability to comply with the proposed protocol assessments or any uncertainty about their ability to give meaningful, informed consent (legal guardian may give consent with patient assent)
7. Concurrent medical conditions representing a contraindication to any of the study medications
8. Grade 3 renal impairment or worse as indicated by eGFR< 60mL/min/1.73m2
9. Clinical evidence of acute liver disease including symptoms of jaundice or right upper quadrant pain or INR >1.8
10. Involvement in another interventional clinical trial within the previous 6 months from baseline
11. Weight <40 kg or >100 kg
12. Male patients and female patients of childbearing potential who are not willing to use appropriate birth control (i.e. double barrier birth control) from enrolment until the follow-up visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Maximum Concentration ( C max) of Trappsol in plasma from patients with Niemann-Pick disease Type C1 by measurement of plasma levels | Pre- infusion then 2 ,4,6,8,8.5,9,10,11 12,16 and 20 hours after the start of the infusions at 1&12 w
  To compare the C max of Trappsol following 2 different dose levels of intravenous Trappsol in patients with NPC-1 disease following single and multiple doses
Time to Maximum Concentration (T max) of Trappsol in plasma from patients with Niemann-Pick disease Type C1 by measurement of plasma levels | Pre- infusion,2 ,4,6,8,8.5,9,10,11 12,16 and 20 hours after the start of the infusions at 1&12 w
  To compare the T max of Trappsol following 2 different dose levels of intravenous Trappsol in patients with NPC-1 disease following single and multiple doses
Volume of Distribution of Trappsol in plasma from patients with Niemann-Pick disease Type C1 by measurement of plasma levels | Pre- infusion,2 ,4,6,8,8.5,9,10,11 12,16 and 20 hours after the start of the infusions at 1&12 w
  To compare the Volume of Distribution of Trappsol following 2 different dose levels of intravenous Trappsol in patients with NPC-1 disease following single and multiple doses
Elimination half-life (T1/2) of Trappsol in plasma from patients with Niemann-Pick disease Type C1 by measurement of plasma levels | Pre- infusion,2 ,4,6,8,8.5,9,10,11 12,16 and 20 hours after the start of the infusions at 1&12 w
  To compare the T1/2 of Trappsol following 2 different doses.

SECONDARY OUTCOMES:
CSF levels of Trappsol | Pre-infusion then 2,4,6,8,12 hours after the first infusion ( w1) and 8h after the start of the last infusion (W12)
  To evaluate HP-β-CD concentrations in CSF following 2 different dose levels of intravenous Trappsol in patients with NPC-1 disease following single and multiple doses
Potential blood biomarkers of NPC1 | Screening, baseline,then at 2,4,8,12 and 14 weeks
  To investigate the effect of 2 different doses of intravenous Trappsol upon peripheral blood biomarkers of NPC-1 disease
Potential CSF biomarkers of NPC1 | Baseline, then at 12 and 14 weeks
  To investigate the effect of 2 different doses of intravenous Trappsol upon biomarkers of NPC-1 disease in CSF
Serum cholesterol precursors and metabolites | Screening, baseline the Days1,3,,5,8,11 and 15 after the first infusion of Trappsol then at d2,3,5,8,11and 15 after the last infusion ( W12)
  To investigate the effect of 2 different doses of intravenous Trappsol in patients with NPC-1 disease upon serum and lymphocytic markers of cholesterol metabolism
Fractionated cholesterol in hepatic tissue | Baseline and 12 weeks
  To investigate the effect of 2 different doses of intravenous Trappsol in patients with NPC-1 disease upon fractionated cholesterol in hepatic tissue
Splenic morphology assessed by qualitative change in ultrasound compared with baseline, NIH total and individual domain severity scores | Baseline then 14 weeks
  To evaluate the effect of 2 different doses of Trappsol upon change in clinical manifestations of NPC-1 disease
Hepatic morphology assessed by qualitative change in ultrasound compared with baseline, NIH total and individual domain severity scores | Baseline then 14 weeks
  To evaluate the effect of 2 different doses of Trappsol upon change in clinical manifestations of NPC-1 disease
Number of patients with treatment-related adverse events as graded by CTCAE criteria ( Version 4.03) | Screening, baseline, days 1, 2-11, weeks 2,4,6,810,12,14 and 18
  Events will be gathered by spontaneous reporting, clinical observation and laboratory tests including auditory tests and auditory evoked potentials to assess hearing

OTHER OUTCOMES:
Hepatic elasticity | Baseline and 14weeks
  To investigate the effect of 2 different doses of intravenous Trappsol upon hepatic elasticity (measured by ultrasound scan) at 14 weeks (after 7 doses) in patients with NPC-1 disease
Filipin signal intensity | Baseline and 12weeks
  To investigate the effect of 2 different doses of intravenous Trappsol on filipin signal intensity (measured in cultured fibroblasts collected by skin biopsy) at 14 weeks (after 7 doses) in patients with NPC-1 disease

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Hastings, MD, Principal Investigator — Oakland CA
Locations (2):
- United States (2):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Atlantic Health System/Morristown Medical Center, Morristown, New Jersey

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Battisti C, Tarugi P, Dotti MT, De Stefano N, Vattimo A, Chierichetti F, Calandra S, Federico A. Adult onset Niemann-Pick type C disease: A clinical, neuroimaging and molecular genetic study. Mov Disord. 2003 Nov;18(11):1405-9. doi: 10.1002/mds.10541. PMID 14639697
- [Background] Coussement W, Van Cauteren H, Vandenberghe J, et al. Toxicological profile of hydroxypropyl Beta-cyclodextrin (HP-Beta-CD) in laboratory animals. In: Minutes of the Fifth International Symposium on cyclodextrins; 28-30 March 1990; Paris, France: Editions de Santé; 1990 p. 522-4.
- [Background] Davidson CD, Ali NF, Micsenyi MC, Stephney G, Renault S, Dobrenis K, Ory DS, Vanier MT, Walkley SU. Chronic cyclodextrin treatment of murine Niemann-Pick C disease ameliorates neuronal cholesterol and glycosphingolipid storage and disease progression. PLoS One. 2009 Sep 11;4(9):e6951. doi: 10.1371/journal.pone.0006951. PMID 19750228
- [Background] Dietschy JM, Turley SD. Control of cholesterol turnover in the mouse. J Biol Chem. 2002 Feb 8;277(6):3801-4. doi: 10.1074/jbc.R100057200. Epub 2001 Dec 3. No abstract available. PMID 11733542
- [Background] Fischer D, Stewart AL, Bloch DA, Lorig K, Laurent D, Holman H. Capturing the patient's view of change as a clinical outcome measure. JAMA. 1999 Sep 22-29;282(12):1157-62. doi: 10.1001/jama.282.12.1157. PMID 10501119
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Giese AK, Mascher H, Grittner U, Eichler S, Kramp G, Lukas J, te Vruchte D, Al Eisa N, Cortina-Borja M, Porter FD, Platt FM, Rolfs A. A novel, highly sensitive and specific biomarker for Niemann-Pick type C1 disease. Orphanet J Rare Dis. 2015 Jun 17;10:78. doi: 10.1186/s13023-015-0274-1. PMID 26082315
- [Background] Gould S, Scott RC. 2-Hydroxypropyl-beta-cyclodextrin (HP-beta-CD): a toxicology review. Food Chem Toxicol. 2005 Oct;43(10):1451-9. doi: 10.1016/j.fct.2005.03.007. Epub 2005 Apr 19. PMID 16018907
- [Background] Greer WL, Dobson MJ, Girouard GS, Byers DM, Riddell DC, Neumann PE. Mutations in NPC1 highlight a conserved NPC1-specific cysteine-rich domain. Am J Hum Genet. 1999 Nov;65(5):1252-60. doi: 10.1086/302620. PMID 10521290
- [Background] Ferraioli G, Parekh P, Levitov AB, Filice C. Shear wave elastography for evaluation of liver fibrosis. J Ultrasound Med. 2014 Feb;33(2):197-203. doi: 10.7863/ultra.33.2.197. PMID 24449721
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] King KA, Gordon-Salant S, Yanjanin N, Zalewski C, Houser A, Porter FD, Brewer CC. Auditory phenotype of Niemann-Pick disease, type C1. Ear Hear. 2014 Jan-Feb;35(1):110-7. doi: 10.1097/AUD.0b013e3182a362b8. PMID 24225652
- [Background] Liu B, Li H, Repa JJ, Turley SD, Dietschy JM. Genetic variations and treatments that affect the lifespan of the NPC1 mouse. J Lipid Res. 2008 Mar;49(3):663-9. doi: 10.1194/jlr.M700525-JLR200. Epub 2007 Dec 12. PMID 18077828
- [Background] Liu B, Turley SD, Burns DK, Miller AM, Repa JJ, Dietschy JM. Reversal of defective lysosomal transport in NPC disease ameliorates liver dysfunction and neurodegeneration in the npc1-/- mouse. Proc Natl Acad Sci U S A. 2009 Feb 17;106(7):2377-82. doi: 10.1073/pnas.0810895106. Epub 2009 Jan 26. PMID 19171898
- [Background] Mattsson N, Zetterberg H, Bianconi S, Yanjanin NM, Fu R, Mansson JE, Porter FD, Blennow K. Miglustat treatment may reduce cerebrospinal fluid levels of the axonal degeneration marker tau in niemann-pick type C. JIMD Rep. 2012;3:45-52. doi: 10.1007/8904_2011_47. Epub 2011 Sep 28. PMID 23430872
- [Background] Naureckiene S, Sleat DE, Lackland H, Fensom A, Vanier MT, Wattiaux R, Jadot M, Lobel P. Identification of HE1 as the second gene of Niemann-Pick C disease. Science. 2000 Dec 22;290(5500):2298-301. doi: 10.1126/science.290.5500.2298. PMID 11125141
- [Background] Neufeld EB, Cooney AM, Pitha J, Dawidowicz EA, Dwyer NK, Pentchev PG, Blanchette-Mackie EJ. Intracellular trafficking of cholesterol monitored with a cyclodextrin. J Biol Chem. 1996 Aug 30;271(35):21604-13. doi: 10.1074/jbc.271.35.21604. PMID 8702948
- [Background] Park WD, O'Brien JF, Lundquist PA, Kraft DL, Vockley CW, Karnes PS, Patterson MC, Snow K. Identification of 58 novel mutations in Niemann-Pick disease type C: correlation with biochemical phenotype and importance of PTC1-like domains in NPC1. Hum Mutat. 2003 Oct;22(4):313-25. doi: 10.1002/humu.10255. PMID 12955717
- [Background] Patterson MC, Vecchio D, Prady H, Abel L, Wraith JE. Miglustat for treatment of Niemann-Pick C disease: a randomised controlled study. Lancet Neurol. 2007 Sep;6(9):765-72. doi: 10.1016/S1474-4422(07)70194-1. PMID 17689147
- [Background] Patterson MC, Hendriksz CJ, Walterfang M, Sedel F, Vanier MT, Wijburg F; NP-C Guidelines Working Group. Recommendations for the diagnosis and management of Niemann-Pick disease type C: an update. Mol Genet Metab. 2012 Jul;106(3):330-44. doi: 10.1016/j.ymgme.2012.03.012. Epub 2012 May 8. PMID 22572546
- [Background] Pontikis CC, Davidson CD, Walkley SU, Platt FM, Begley DJ. Cyclodextrin alleviates neuronal storage of cholesterol in Niemann-Pick C disease without evidence of detectable blood-brain barrier permeability. J Inherit Metab Dis. 2013 May;36(3):491-8. doi: 10.1007/s10545-012-9583-x. Epub 2013 Feb 15. PMID 23412751
- [Background] Ramirez CM, Liu B, Aqul A, Taylor AM, Repa JJ, Turley SD, Dietschy JM. Quantitative role of LAL, NPC2, and NPC1 in lysosomal cholesterol processing defined by genetic and pharmacological manipulations. J Lipid Res. 2011 Apr;52(4):688-98. doi: 10.1194/jlr.M013789. Epub 2011 Feb 2. PMID 21289032
- [Background] Schicks J, Muller Vom Hagen J, Bauer P, Beck-Wodl S, Biskup S, Krageloh-Mann I, Schols L, Synofzik M. Niemann-Pick type C is frequent in adult ataxia with cognitive decline and vertical gaze palsy. Neurology. 2013 Mar 19;80(12):1169-70. doi: 10.1212/WNL.0b013e31828869f9. Epub 2013 Feb 20. No abstract available. PMID 23427322
- [Background] Schmitz-Hubsch T, du Montcel ST, Baliko L, Berciano J, Boesch S, Depondt C, Giunti P, Globas C, Infante J, Kang JS, Kremer B, Mariotti C, Melegh B, Pandolfo M, Rakowicz M, Ribai P, Rola R, Schols L, Szymanski S, van de Warrenburg BP, Durr A, Klockgether T, Fancellu R. Scale for the assessment and rating of ataxia: development of a new clinical scale. Neurology. 2006 Jun 13;66(11):1717-20. doi: 10.1212/01.wnl.0000219042.60538.92. PMID 16769946
- [Background] Sevin M, Lesca G, Baumann N, Millat G, Lyon-Caen O, Vanier MT, Sedel F. The adult form of Niemann-Pick disease type C. Brain. 2007 Jan;130(Pt 1):120-33. doi: 10.1093/brain/awl260. Epub 2006 Sep 26. PMID 17003072
- [Background] Tangemo C, Weber D, Theiss S, Mengel E, Runz H. Niemann-Pick Type C disease: characterizing lipid levels in patients with variant lysosomal cholesterol storage. J Lipid Res. 2011 Apr;52(4):813-25. doi: 10.1194/jlr.P013524. Epub 2011 Jan 17. PMID 21245028
- [Background] te Vruchte D, Speak AO, Wallom KL, Al Eisa N, Smith DA, Hendriksz CJ, Simmons L, Lachmann RH, Cousins A, Hartung R, Mengel E, Runz H, Beck M, Amraoui Y, Imrie J, Jacklin E, Riddick K, Yanjanin NM, Wassif CA, Rolfs A, Rimmele F, Wright N, Taylor C, Ramaswami U, Cox TM, Hastings C, Jiang X, Sidhu R, Ory DS, Arias B, Jeyakumar M, Sillence DJ, Wraith JE, Porter FD, Cortina-Borja M, Platt FM. Relative acidic compartment volume as a lysosomal storage disorder-associated biomarker. J Clin Invest. 2014 Mar;124(3):1320-8. doi: 10.1172/JCI72835. PMID 24487591
- [Background] Trendelenburg G, Vanier MT, Maza S, Millat G, Bohner G, Munz DL, Zschenderlein R. Niemann-Pick type C disease in a 68-year-old patient. J Neurol Neurosurg Psychiatry. 2006 Aug;77(8):997-8. doi: 10.1136/jnnp.2005.086785. No abstract available. PMID 16844962
- [Background] Vance JE. Dysregulation of cholesterol balance in the brain: contribution to neurodegenerative diseases. Dis Model Mech. 2012 Nov;5(6):746-55. doi: 10.1242/dmm.010124. Epub 2012 Oct 12. PMID 23065638
- [Background] Vanier MT. Niemann-Pick disease type C. Orphanet J Rare Dis. 2010 Jun 3;5:16. doi: 10.1186/1750-1172-5-16. PMID 20525256
- [Background] Vite CH, Bagel JH, Swain GP, Prociuk M, Sikora TU, Stein VM, O'Donnell P, Ruane T, Ward S, Crooks A, Li S, Mauldin E, Stellar S, De Meulder M, Kao ML, Ory DS, Davidson C, Vanier MT, Walkley SU. Intracisternal cyclodextrin prevents cerebellar dysfunction and Purkinje cell death in feline Niemann-Pick type C1 disease. Sci Transl Med. 2015 Feb 25;7(276):276ra26. doi: 10.1126/scitranslmed.3010101. PMID 25717099
- [Background] Welford RW, Garzotti M, Marques Lourenco C, Mengel E, Marquardt T, Reunert J, Amraoui Y, Kolb SA, Morand O, Groenen P. Plasma lysosphingomyelin demonstrates great potential as a diagnostic biomarker for Niemann-Pick disease type C in a retrospective study. PLoS One. 2014 Dec 5;9(12):e114669. doi: 10.1371/journal.pone.0114669. eCollection 2014. PMID 25479233
- [Derived] Hastings C, Liu B, Hurst B, Cox GF, Hrynkow S. Intravenous 2-hydroxypropyl-beta-cyclodextrin (Trappsol(R) Cyclo) demonstrates biological activity and impacts cholesterol metabolism in the central nervous system and peripheral tissues in adult subjects with Niemann-Pick Disease Type C1: Results of a phase 1 trial. Mol Genet Metab. 2022 Dec;137(4):309-319. doi: 10.1016/j.ymgme.2022.10.004. Epub 2022 Oct 17. PMID 36279795